CLINICAL TRIAL: NCT03368599
Title: The Effect of Endobronchial Intubation of Double-lumen Tube on Post-operative Sore Throat, Hoarseness and Airway Injuries: A Comparison Between Conventional and Fiberoptic Bronchoscope-guided Intubation
Brief Title: Endobronchial Intubation of Double-lumen Tube: Conventional Method vs Fiberoptic Bronchoscope Guide Method
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Jin-Woo Park, Assistant Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: B-1711-432-005
Record Dates: First submitted 2017-12-01; First posted 2017-12-11 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Intubation, Intratracheal; Postoperative Complications; Sore Throat; Hoarseness; Soft Tissue Injuries; Thoracic Surgery
MeSH Terms: conditions — Postoperative Complications; Pharyngitis; Hoarseness; Soft Tissue Injuries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bronchoscope guide group (Experimental): DLT is advanced into the main bronchus through the guide of fiberoptic bronchoscope (Bronchoscope guided advancement).
  Interventions: Procedure: Bronchoscope guided advancement
- Conventional group (Active Comparator): DLT is advanced blindly to the main bronchus level (Conventional advancement).
  Interventions: Procedure: Conventional advancement

INTERVENTIONS:
Procedure: Bronchoscope guided advancement — During the anesthetic induction for thoracic surgery, Lt. DLT is intubated using the bronchoscope-guided method. The method is as follows.
  1. Lt. DLT is intubated through vocal cord using the direct laryngoscopy.
  2. Pass the fiberoptic bronschoscope through a bronchial lumen of Lt. DLT.
  3. Secure the pathway into the Lt. main bronchus by advancing the bronchoscope into the Lt. main bronchus.
  4. Lt. DLT can be advanced through the guide of the bronchoscope into Lt. main bronchus.
  5. After the advancement, the position of Lt. DLT can be confirmed using the fiberoptic bronchoscope. If necessary, the depth and direction of Lt. DLT should be modified.
  Arms: Bronchoscope guide group
Procedure: Conventional advancement — During the anesthetic induction for thoracic surgery, Lt. DLT is intubated using the conventional method. The method is as follows.
  1. Lt. DLT is intubated through vocal cord using the direct laryngoscopy.
  2. Rotate Lt. DLT 90 degrees to the left side.
  3. Advance Lt. DLT blindly to main bronchus level.
  4. After the advancement, the position of Lt. DLT can be confirmed using the fiberoptic bronchoscope. If necessary, the depth and direction of Lt. DLT should be modified.
  Arms: Conventional group

SUMMARY:
Double lumen tube (DLT) needs to be intubated to isolate ventilations of left and right lungs for thoracic surgery. Post-operative sore throat and hoarseness are more frequent with DLT intubation than with single one. Which is may because DLT is relatively thicker, harder, sideway curved and therefore more likely to damage the vocal cord or trachea during intubation, and advanced deeper to the carina and main bronchus level. In the conventional method of intubation, DLT is rotated 90 degrees and advanced blindly to the main bronchus level after DLT is intubated through vocal cord using the direct laryngoscopy. After the blind advancement, the sufficient tube position needs to be gained and confirmed with the fiberoptic bronchoscope. In the bronchoscope guide method, after DLT is intubated through vocal cord using the direct laryngoscopy, the pathway into the targeted main bronchus is secured using the fiberoptic bronchoscope which is passed through a bronchial lumen of DLT. And then DLT can be advanced through the guide of the bronchoscope. In this study, we intend to compare post-operative sore throat, hoarseness and airway injury between the two methods. We hypothesize that the bronchoscope guide method can reduce the post-operative complications and airway injury because surrounding tissues of the airway can be less irritated by DLT intubation in the guide method than in a conventional.

For a constant guide effect, we use fiberoptic bronchoscopes with same outer diameter (4.1 mm) which can pass through a bronchial lumen of 37 and 39 Fr Lt. DLT and cannot pass through 35 Fr or smaller Lt. DLTs.

<Lt. DLT size selection>

* male: ≥160 cm, 39 French; < 160 cm, 37 French
* female: ≥160 cm, 37 French; < 160 cm, contraindication

ELIGIBILITY:
Inclusion Criteria:

* ASA (American Society of Anesthesiologists) class I - III
* Elective thoracic surgery
* Left-sided DLT intubation for one-lung ventilation

Exclusion Criteria:

* Female, height < 160 cm
* Pre-existing sore throat, hoarseness or airway injury
* Duration of surgery > 6 h
* Upper respiratory tract infection
* Cervical spine diseases
* Presence of tracheostomy
* Pharyngeal neoplasm or abscess which can induce mechanical airway obstruction
* Mallampati score 4
* Obesity (BMI ≥ 35 kg/m2)
* Obstructive sleep apnea (OSA)
* Craniofacial anomaly
* Cormack grade 3b or 4
* History or high risk of difficult intubation / difficult mask ventilation
* Patients whom the direct laryngoscopy cannot be used for, because of weak teeth or small mouth opening
* Patients who refuse to participate in the study or from whom receive informed consent cannot be received.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2019-01-30 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Post-operative sore throat (24 h) | 24 hour after tracheal extubation
  The degree of throat pain (Visual Analogue Scale (VAS); 0, no pain; 10, most

SECONDARY OUTCOMES:
Resistance against DLT passage through vocal cord | Intraoperative
  none/mild/severe
Resistance against DLT advancement | Intraoperative
  none/mild/severe
Intubation time | Intraoperative
  stop of initial mask ventilation - intubation through vocal cord
The number of attempts for intubation | Intraoperative
  The number of attempts for intubation through vocal cord
The number of right misplacement of Lt. DLT | Intraoperative
  The number of right misplacement of Lt. DLT confirmed using the fiberoptic bronchoscope after the advancement
Time for DLT positioning: stop of initial mask ventilation - success of the 1st fine DLT positioning | Intraoperative
  Time for DLT positioning: stop of initial mask ventilation - success of the 1st fine DLT positioning into Lt. main bronchus
Heart rate | Intraoperative
  Heart rate Just before Lt. DLT intubation / 2 min after success of the 1st fine DLT positioning
Mean arterial pressure | Intraoperative
  Mean arterial pressure Just before Lt. DLT intubation / 2 min after success of the 1st fine DLT positioning
IV PCA | At 24 hours after the extubation
  Fentanyl usage with PCA
Airway injury (Lt. main bronhcus, carina, trachea) | Intraoperative
  When spontaneous breathing of the patient starts after the thoracic surgery
Airway injury (vocal cord) | Intraoperative
  When spontaneous breathing of the patient starts after the thoracic surgery
Post-operative sore throat (1 h) | 24 hours after tracheal extubation
  The degree of throat pain (Visual Analogue Scale (VAS); 0, no pain; 10, most pain) after tracheal extubation
Post-operative hoarseness (1 h) | 1 hour after tracheal extubation
  The incidence of hoarseness after tracheal extubation
Post-operative hoarseness (24 h) | 24 hour after tracheal extubation
  The incidence of hoarseness after tracheal extubation
Oral dryness | 24 hours after tracheal extubation
  The incidence of oral dryness
Dysphagia | 24 hours after tracheal extubation
  The incidence of dysphagia

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Woo Park, MD, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Christensen AM, Willemoes-Larsen H, Lundby L, Jakobsen KB. Postoperative throat complaints after tracheal intubation. Br J Anaesth. 1994 Dec;73(6):786-7. doi: 10.1093/bja/73.6.786. PMID 7880666
- [Background] McHardy FE, Chung F. Postoperative sore throat: cause, prevention and treatment. Anaesthesia. 1999 May;54(5):444-53. doi: 10.1046/j.1365-2044.1999.00780.x. PMID 10995141
- [Background] Chang JE, Min SW, Kim CS, Han SH, Kwon YS, Hwang JY. Effect of prophylactic benzydamine hydrochloride on postoperative sore throat and hoarseness after tracheal intubation using a double-lumen endobronchial tube: a randomized controlled trial. Can J Anaesth. 2015 Oct;62(10):1097-103. doi: 10.1007/s12630-015-0432-x. Epub 2015 Jul 7. PMID 26149601
- [Background] Park SH, Han SH, Do SH, Kim JW, Rhee KY, Kim JH. Prophylactic dexamethasone decreases the incidence of sore throat and hoarseness after tracheal extubation with a double-lumen endobronchial tube. Anesth Analg. 2008 Dec;107(6):1814-8. doi: 10.1213/ane.0b013e318185d093. PMID 19020122
- [Result] Seo JH, Cho CW, Hong DM, Jeon Y, Bahk JH. The effects of thermal softening of double-lumen endobronchial tubes on postoperative sore throat, hoarseness and vocal cord injuries: a prospective double-blind randomized trial. Br J Anaesth. 2016 Feb;116(2):282-8. doi: 10.1093/bja/aev414. PMID 26787799
- [Result] Cheong KF, Koh KF. Placement of left-sided double-lumen endobronchial tubes: comparison of clinical and fibreoptic-guided placement. Br J Anaesth. 1999 Jun;82(6):920-1. doi: 10.1093/bja/82.6.920. PMID 10562789
- [Result] Knoll H, Ziegeler S, Schreiber JU, Buchinger H, Bialas P, Semyonov K, Graeter T, Mencke T. Airway injuries after one-lung ventilation: a comparison between double-lumen tube and endobronchial blocker: a randomized, prospective, controlled trial. Anesthesiology. 2006 Sep;105(3):471-7. doi: 10.1097/00000542-200609000-00009. PMID 16931978
- [Derived] Park JW, Jo JH, Park JH, Bae YK, Park SJ, Cho SW, Han SH, Kim JH. Comparison of conventional and fibreoptic-guided advance of left-sided double-lumen tube during endobronchial intubation: A randomised controlled trial. Eur J Anaesthesiol. 2020 Jun;37(6):466-473. doi: 10.1097/EJA.0000000000001216. PMID 32332265